CLINICAL TRIAL: NCT03095651
Title: A Study to Assess the Safety, Pharmacokinetics and Pharmacodynamic Effect of MK-5160 in Subjects With Type 1 and Type 2 Diabetes Mellitus
Brief Title: Multiple Ascending Dose Study of MK-5160 in Participants With Type 1 and Type 2 Diabetes Mellitus (MK-5160-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5160-002; MK-5160-002 (Other: Merck protocol number)
Record Dates: First submitted 2017-03-27; First posted 2017-03-29 (Actual); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- T1DM MK-5160 16 nmol/kg (Experimental): Participants with T1DM received MK-5160, 16 nmol/kg, and placebo to glargine daily for 12 days. Dextrose was administered as needed to maintain blood sugar.
  Interventions: Biological: MK-5160 16 nmol/kg; Biological: Placebo to Glargine; Drug: Dextrose
- T1DM MK-5160 32 nmol/kg (Experimental): Participants with T1DM received MK-5160, 32 nmol/kg, and placebo to glargine daily for 12 days. Dextrose was administered as needed to maintain blood sugar.
  Interventions: Biological: MK-5160 32 nmol/kg; Biological: Placebo to Glargine; Drug: Dextrose
- T1DM MK-5160 64 nmol/kg (Experimental): Participants with T1DM received MK-5160 64 nmol/kg, and placebo to glargine daily for 12 days. Dextrose was administered as needed to maintain blood sugar.
  Interventions: Biological: MK-5160 64 nmol/kg; Biological: Placebo to Glargine; Drug: Dextrose
- T1DM Glargine 0.4 U/kg (Active Comparator): Participants with T1DM received Glargine 0.4 U/kg and placebo to MK-5160 daily for 12 days. Dextrose was administered as needed to maintain blood sugar.
  Interventions: Biological: Glargine 0.4 U/kg; Biological: Placebo to MK-5160; Drug: Dextrose
- T2DM MK-5160 16 nmol/kg (Experimental): Participants with T2DM received MK-5160 16 nmol/kg, and placebo to glargine daily for 12 days. Dextrose was administered as needed to maintain blood sugar.
  Interventions: Biological: MK-5160 16 nmol/kg; Biological: Placebo to Glargine; Drug: Dextrose
- T2DM MK-5160 32 nmol/kg (Experimental): Participants with T2DM received MK-5160 32 nmol/kg, and placebo to glargine daily for 12 days. Dextrose was administered as needed to maintain blood sugar.
  Interventions: Biological: MK-5160 32 nmol/kg; Biological: Placebo to Glargine; Drug: Dextrose
- T2DM MK-5160 64 nmol/kg (Experimental): Participants with T2DM received MK-5160 64 nmol/kg, and placebo to glargine daily for 12 days. Dextrose was administered as needed to maintain blood sugar.
  Interventions: Biological: MK-5160 64 nmol/kg; Biological: Placebo to Glargine; Drug: Dextrose
- T2DM Glargine 0.6 U/kg (Active Comparator): Participants with T2DM received Glargine 0.6 U/kg and placebo to MK-5160 daily for 12 days. Dextrose was administered as needed to maintain blood sugar.
  Interventions: Biological: Placebo to MK-5160; Drug: Dextrose; Biological: Glargine 0.6 U/kg

INTERVENTIONS:
Biological: MK-5160 16 nmol/kg — MK-5160 16 nmol/kg, subcutaneous injection administered daily for 12 days
  Arms: T1DM MK-5160 16 nmol/kg; T2DM MK-5160 16 nmol/kg
Biological: MK-5160 32 nmol/kg — MK-5160 32 nmol/kg, subcutaneous injection administered daily for 12 days
  Arms: T1DM MK-5160 32 nmol/kg; T2DM MK-5160 32 nmol/kg
Biological: MK-5160 64 nmol/kg — MK-5160 64 nmol/kg, subcutaneous injection administered daily for 12 days
  Arms: T1DM MK-5160 64 nmol/kg; T2DM MK-5160 64 nmol/kg
Biological: Glargine 0.4 U/kg — Glargine 0.4 U/kg, subcutaneous injection administered daily for 12 days
  Arms: T1DM Glargine 0.4 U/kg
Biological: Placebo to Glargine — Placebo to glargine, subcutaneous injection administered daily for 12 days
  Arms: T1DM MK-5160 16 nmol/kg; T1DM MK-5160 32 nmol/kg; T1DM MK-5160 64 nmol/kg; T2DM MK-5160 16 nmol/kg; T2DM MK-5160 32 nmol/kg; T2DM MK-5160 64 nmol/kg
Biological: Placebo to MK-5160 — Placebo to MK-5160, subcutaneous injection administered daily for 12 days
  Arms: T1DM Glargine 0.4 U/kg; T2DM Glargine 0.6 U/kg
Drug: Dextrose — 20% solution of dextrose; adjusted to maintain the various glycemic levels at 100 mg/dL given as a continuous intravenous infusion for 6-30 hours.
Biological: Glargine 0.6 U/kg — Glargine 0.6 U/kg, subcutaneous injection administered daily for 12 days
  Arms: T2DM Glargine 0.6 U/kg

SUMMARY:
This is a randomized, active- and placebo-controlled, double-blind trial of MK-5160 in participants with Type 1 diabetes mellitus (T1DM) and Type 2 diabetes mellitus (T2DM). This is a two-part trial, with three panels per part. T1DM (Part 1) and T2DM (Part 2) participants will be given daily fixed doses of MK-5160 in three predefined, increasing doses in each panel, or glargine (active comparator). The primary hypothesis of the trial is that at a dose with sufficient safety, the mean steady-state maximum level of glucose infusion rate (GIRmax) after MK-5160 administration in both T1DM and T2DM participants is between 1.5 and 4.5 mg/kg/min.

ELIGIBILITY:
Inclusion Criteria:

* For Part 1 (T1DM):
* Be male, or female of non-childbearing potential. A female of non-childbearing potential defined as a female who is postmenopausal without menses for at least 1 year and has a follicle stimulating hormone (FSH) value in the postmenopausal range upon pretrial (screening) evaluation OR a female who is status post hysterectomy, oophorectomy or tubal ligation.
* Be judged to be in good health
* Have a diagnosis of T1DM as defined by standard diagnostic criteria for ≥12 months at time study participation
* Be on stable doses of basal insulin over the 2-week period prior to screening and over the 2 weeks prior to dosing.
* Have a total daily insulin requirement (basal plus prandial) of ≤ 1.2 units/kg.
* Have a hemoglobin A1C (HbA1c) ≤10% at the time of study participation.
* Have a Body Mass Index (BMI) ≥18.5 kg/m^2 and ≤ 32 kg/m^2. BMI = mass (kg)/height (m)^2
* Be a non-smoker or smoker who uses no more than 5 cigarettes or equivalent (e.g., e-cigarettes) per day over the prior 3 month period also may be enrolled (at the discretion of the investigator). The subject must agree to follow the smoking restrictions defined by the clinical research unit (CRU).
* For Part 2 (T2DM):
* Be male, or female of non-childbearing potential. A female of non-childbearing potential defined as a female who is postmenopausal without menses for at least 1 year and has a FSH value in the postmenopausal range upon pretrial (screening) evaluation OR a female who is status post hysterectomy, oophorectomy or tubal ligation.
* Be judged to be in good health
* Have a diagnosis of T2DM as defined by standard diagnostic criteria for ≥12 month at time of study participation.
* T2DM participants are not required to have been on insulin. If on insulin, participants should have a total daily insulin requirement of ≤ 1.2 units/kg, and have been on stable doses of basal insulin over the 2-week period prior to screening and over the 2 weeks prior to dosing.
* Meet one of the following criteria:

  1. Be on no anti-hyperglycemic agent (AHA), or on metformin monotherapy or metformin plus a dipeptidyl peptidase-4 (DPP4) inhibitor at stable doses for at least 8 weeks prior to screening, with a screening HbA1C ≥7.0 and ≤10.0%.
  2. Be on either a sulfonylurea (e.g. glyburide) or an alpha-glucosidase inhibitors (e.g., acarbose) alone or in combination with metformin at stable doses for at least 8 weeks prior to screening with a screening HbA1C ≥7.0 and ≤9.0%. Participants on these medications must be willing to stop the sulfonylurea or alpha-glucosidase inhibitor after screening once they qualify for study participation.
* Have a BMI ≥18.5 kg/m^2 and ≤ 35.0 kg/m^2 BMI = mass (kg)/height (m)^2
* May be on selected standard medications for T2DM, including alpha-glucosidase inhibitors (e.g., acarbose), sulfonylureas (e.g. glyburide), DPP-4 inhibitors, and metformin. Participants on alpha-glucosidase inhibitors and/or sulfonylureas must stop these medications for at least one week prior to checking into the site and for the duration of the trial through the last dose of MK-5160/glargine. Participants on metformin or DPP-4 inhibitors may continue on their home dose for the duration of the trial. Participants on SGLT2 inhibitors (gliflozins), thiazolidinediones or GLP-1 agonists are excluded.
* Be a nonsmoker or smoker who uses no greater than 5 cigarettes or equivalent (e.g., e-cigarettes) daily over the prior 3 month period. Participants must agree to follow the smoking restrictions defined by the CRU.

Exclusion Criteria:

* For Part 1 (T1DM) and Part 2 (T2DM):
* Is under the age of legal consent
* Is mentally or legally incapacitated, has significant emotional problems at the time of pretrial (screening) visit or expected during the conduct of the trial or has a history of clinically significant psychiatric disorder of the last 5 years. Participants who have had situational depression may be enrolled in the trial at the discretion of the investigator.
* Has a history of clinically significant endocrine (excluding diabetes mellitus), gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases. Participants with a history of uncomplicated kidney stones, as defined as spontaneous passage and no recurrence in the last 5 years, or childhood asthma may be enrolled in the trial at the discretion of the investigator.
* Has a history of cancer (malignancy) Exceptions: (1) Participants with adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix may participate in the trial; (2) Participants with other malignancies which have been successfully treated ≥10 years prior to the pretrial visit
* Has a history of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e. systemic allergic reaction) to prescription or non-prescription drugs or food.
* Is positive for hepatitis B surface antigen, hepatitis C antibodies or HIV at Screening.
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pretrial visit.
* Has participated in another investigational trial within 4 weeks (or 5 half-lives), whichever is greater, prior to the pretrial visit.
* Is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of trial drug, throughout the trial (including washout intervals between treatment periods), until the post-trial visit. Certain medications, such as antihypertensives and aspirin, are permitted.
* Consumes greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day.
* Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy-drinks, or other caffeinated beverages per day.
* Is a regular user of cannabis or any illicit drugs, or has a history of drug (including alcohol) abuse within approximately 6 months.
* Has the diagnosis of hypoglycemia unawareness, or has had one or more severe hypoglycemic episodes associated with hypoglycemic seizures, comas or unconsciousness within 6 months prior to dosing.
* Has used systemic (intravenous, oral, inhaled) glucocorticoids within 3 months of screening or is anticipated to require treatment with systemic glucocorticoids during study participation.
* Has other major medical problems requiring medication (i.e., history of myocardial infarction, hypercholesterolemia). Participants on aspirin as prophylaxis may be enrolled, provided there is no history of MI or other thromboembolic event, or a history of coronary atherosclerosis.
* Has a known history of celiac disease or significant food allergy, at the discretion of the Investigator and Sponsor.
* Has a history of hypersensitivity to pharmacologic insulins or to any of the inactive ingredients in regular human insulin, or to any E.coli-derived drug product.
* For Part 1 (T1DM) Only:
* Has a history of diabetic ketoacidosis in the last 12 months.
* For Part 2 (T2DM) Only
* Has been treated with a sodium/glucose cotransporter 2 (SGLT2) inhibitor (gliflozins), thiazolidinedione or Glucagon-like peptide-1 (GLP-1) receptor agonist within the past three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- ProSciento Inc. ( Site 0001), Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were randomized to the T1DM (Type 1 Diabetes Mellitus) MK-5160 64 nmol/kg arm or the T2DM (Type 2 Diabetes Mellitus) MK-5160 16 nmol/kg arm.
Period: Overall Study
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Started | 6 | 6 | 0 | 4 | 0 | 7 | 6 | 4
Completed | 5 | 5 | 0 | 3 | 0 | 6 | 6 | 4
Not Completed | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were randomized to the T1DM MK-5160 64 nmol/kg arm or the T2DM MK-5160 16 nmol/kg arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg | Total
Number analyzed (Participants) | 6 | 6 | 0 | 4 | 0 | 7 | 6 | 4 | 33
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 64 years | 6 | 6 | 0 | 4 | 0 | 6 | 6 | 4 | 32
  From 65 to 84 years | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 6
  Male | 5 | 6 | 0 | 4 | 0 | 3 | 6 | 3 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 6 | 5 | 0 | 4 | 0 | 7 | 6 | 4 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 33 days
Population: All participants who received at least one dose of study drug. No participants were randomized to the T1DM MK-5160 64 nmol/kg arm or the T2DM MK-5160 16 nmol/kg arm.
Measure: Count of Participants; unit: Participants
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 6 | 6 | 0 | 4 | 0 | 7 | 6 | 4
Participants | 6 | 6 | 0 | 4 | 0 | 7 | 6 | 4

2. Primary Outcome: Number of Participants Discontinuing Study Drug Due to an AE
Description: as for outcome 1
Time Frame: Up to 12 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 6 | 6 | 0 | 4 | 0 | 7 | 6 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Maximal Glucose Infusion Rate
Description: Maximal glucose infusion rate required to maintain target glucose levels in a euglycemic clamp setting (GIRmax) at steady state (Day 12) following administration of study drug. In cases where the lower bound of the CI was negative, the lower confidence limit was truncated at zero. In these cases, the confidence intervals are 97.5% CIs.
Time Frame: Up to 24 hours post-dose on Day 12
Population: All participants that received study drug, had no major protocol violations, and had GIRmax values available on Day 12. No participants were randomized to the T1DM MK-5160 64 nmol/kg arm or the T2DM MK-5160 16 nmol/kg arm.
Measure: Mean (95% Confidence Interval); unit: mg/kg/min
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 6 | 6 | 0 | 4 | 0 | 6 | 6 | 4
mg/kg/min | 2.15 [1.04 to 3.25] | 2.86 [1.80 to 3.92] |  | 2.56 [1.26 to 3.86] |  | 1.98 [1.03 to 2.93] | 2.15 [1.15 to 3.14] | 3.25 [2.03 to 4.47]

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-5160
Description: Cmax of MK-5160 following multiple dose administration of study drug. Glargine data are presented in the following outcome measure.
Time Frame: Day 1 clamp: -15 min. (predose), 10, 30 min., 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours following start of injection (FSOI). Day 12: -15 min (predose), 10, 30 min., 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, and 168 hours FSOI.
Population: All participants that received MK-5160, had no major protocol violations, and had Cmax values available on Day 1 and Day 12. No participants were randomized to the T1DM MK-5160 64 nmol/kg or T2DM MK-5160 16 nmol/kg arms. One participant in the T2DM MK-5160 32 nmol/kg arm withdrew consent after receiving a single dose of study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 7 | 6 | 0
nM
  Day 1 | 0.76 [0.59 to 0.97] | 1.58 [0.99 to 2.53] |  |  |  | 1.33 [0.97 to 1.82] | 1.91 [1.22 to 2.99] |
  Day 12: number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 6 | 6 | 0
  Day 12 | 2.33 [1.75 to 3.10] | 5.38 [3.33 to 8.69] |  |  |  | 3.85 [2.94 to 5.05] | 9.03 [7.73 to 10.55] |

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Glargine
Description: Cmax of glargine following multiple dose administration of study drug. MK-5160 data are presented in the preceding outcome measure.
Time Frame: Day 1 clamp: -15 min. (predose), 10, 30 min., 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours FSOI. Day 12: -15 min (predose), 10, 30 min., 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, and 168 hours FSOI.
Population: All participants that received glargine, had no major protocol violations, and had Cmax values available on Day 1 and Day 12.
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 4
pmol/L
  Day 1 |  |  |  | 17.26 [13.12 to 22.70] |  |  |  | 18.97 [5.29 to 68.00]
  Day 12 |  |  |  | 20.28 [10.74 to 38.28] |  |  |  | 34.18 [12.73 to 91.76]

6. Secondary Outcome: Day 12 to Day 1 Accumulation Ratio of Cmax
Description: Day 12 to Day 1 accumulation ratio (AR) of Cmax of MK-5160 and glargine following multiple dose administration of study drug. Geometric mean accumulation ratio = Day 12 Cmax/Day 1 Cmax.
Time Frame: as for outcome 5
Population: Participants with Cmax measurements on Day 1 and Day 12. No participants were randomized to the T1DM MK-5160 64 nmol/kg arm or the T2DM MK-5160 16 nmol/kg arm.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 6 | 6 | 0 | 4 | 0 | 7 | 6 | 4
Ratio | 3.08 [2.37 to 4.00] | 3.40 [2.11 to 5.48] |  | 1.17 [0.80 to 1.74] |  | 2.89 [2.13 to 3.93] | 4.72 [3.46 to 6.44] | 1.80 [0.65 to 5.01]

7. Secondary Outcome: Steady State Plasma Concentration (Css) of MK-5160
Description: Css of MK-5160 is the amount of MK-5160 in a given volume of plasma at the time a "steady state" has been achieved, and rates of MK-5160 administration and MK-5160 elimination are equal. Glargine data are presented in the following outcome measure.
Time Frame: Day 12: -15 min (predose), 10, 30 min., 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, and 168 hours FSOI.
Population: All participants that received MK-5160, had no major protocol violations, and had Css values available on Day 12. No participants were randomized to the T1DM MK-5160 64 nmol/kg arm or the T2DM MK-5160 16 nmol/kg arm.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 6 | 6 | 0
nM | 1.79 [1.32 to 2.42] | 4.40 [2.55 to 7.57] |  |  |  | 2.64 [1.95 to 3.56] | 6.15 [5.73 to 6.61] |

8. Secondary Outcome: Steady State Plasma Concentration (Css) of Glargine
Description: Css of glargine is the amount of glargine in a given volume of plasma at the time a "steady state" has been achieved, and rates of glargine administration and glargine elimination are equal. MK-5160 data are presented in the preceding outcome measure.
Time Frame: Day 12: -15 min (predose), 10, 30 min., 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, and 168 hours FSOI.
Population: All participants that received glargine, had no major protocol violations, and had Css values available on Day 12.
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 4
pmol/L |  |  |  | 9.99 [3.32 to 30.12] |  |  |  | 14.72 [3.45 to 62.74]

9. Secondary Outcome: Plasma Concentration/Time (AUC0-24) of MK-5160
Description: Area Under the Plasma Concentration/Time Curve for MK-5160 from Time 0 to 24 hours (AUC0-24) is a measure of the total amount of MK-5160 in the plasma from the dose administration to 24 hours. Glargine data are presented in the following outcome measure.
Time Frame: Day 1 clamp: -15 min. (predose), 10, 30 min., 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours FSOI. Day 12: -15 min (predose), 10, 30 min., 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours FSOI.
Population: All participants that received MK-5160, had no major protocol violations, and had AUC0-24 values available on Day 1 and Day 12. No participants were randomized to the T1DM MK-5160 64 nmol/kg or T2DM MK-5160 16 nmol/kg arms. One participant in the T2DM MK-5160 32 nmol/kg arm withdrew consent after receiving a single dose of study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*nM
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 7 | 6 | 0
hr*nM
  Day 1 | 9.79 [7.80 to 12.29] | 26.39 [15.21 to 45.76] |  |  |  | 17.44 [10.88 to 27.94] | 25.32 [16.61 to 38.59] |
  Day 12: number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 6 | 6 | 0
  Day 12 | 42.90 [31.64 to 58.17] | 105.5 [61.30 to 181.7] |  |  |  | 63.29 [46.83 to 85.52] | 147.7 [137.5 to 158.6] |

10. Secondary Outcome: Plasma Concentration/Time (AUC0-24) of Glargine
Description: AUC0-24 is a measure of the total amount of glargine in the plasma from the dose administration to 24 hours. MK-5160 data are presented in the preceding outcome measure.
Time Frame: as for outcome 9
Population: All participants that received glargine, had no major protocol violations, and had AUC0-24 values available on Day 1 and Day 12.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*pmol/L
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 4
hr*pmol/L
  Day 1 |  |  |  | 193.6 [96.81 to 387.2] |  |  |  | 149.6 [13.94 to 1605]
  Day 12 |  |  |  | 239.8 [79.57 to 722.9] |  |  |  | 353.3 [82.90 to 1506]

11. Secondary Outcome: Day 12 to Day 1 Accumulation Ratio of AUC0-24.
Description: Day 12 to Day 1 Accumulation Ratio (AR) of the AUC0-24 of study drug (MK-5160 or glargine). Geometric mean accumulation ratio = Day 12 AUC0-24/Day 1 AUC0-24
Time Frame: as for outcome 9
Population: Participants with AUC0-24 measurements on Day 1 and Day 12. No participants were randomized to the T1DM MK-5160 64 nmol/kg arm or the T2DM MK-5160 16 nmol/kg arm.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 6 | 6 | 0 | 4 | 0 | 7 | 6 | 4
Ratio | 4.38 [3.34 to 5.74] | 4.00 [2.30 to 6.94] |  | 1.24 [0.77 to 1.99] |  | 3.63 [2.37 to 5.56] | 5.83 [4.30 to 7.91] | 2.36 [0.41 to 13.74]

12. Secondary Outcome: Plasma Clearance
Description: Plasma Clearance (CL) of study drug is the volume of plasma cleared of study drug per unit time.
Time Frame: Day 12: -15 min (predose), 10, 30 min., 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, and 168 hours FSOI.
Population: All participants that received study drug, had no major protocol violations, and had CL values available on Day 12. No participants were randomized to the T1DM MK-5160 64 nmol/kg arm or the T2DM MK-5160 16 nmol/kg arm.
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr/kg
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 6 | 6 | 0 | 4 | 0 | 6 | 6 | 4
L/hr/kg | 0.37 [0.28 to 0.51] | 0.30 [0.18 to 0.52] |  | 10.01 [3.32 to 30.16] |  | 0.51 [0.37 to 0.68] | 0.43 [0.40 to 0.47] | 10.19 [2.39 to 43.43]

13. Secondary Outcome: Time to Maximum Plasma Concentration
Description: Time to reach the maximum plasma concentration (Tmax) of study drug after the dose is given.
Time Frame: as for outcome 5
Population: All participants that received study drug, had no major protocol violations, and had Tmax values available on Day 1 and Day 12. No participants were randomized to the T1DM MK-5160 64 nmol/kg arm or the T2DM MK-5160 16 nmol/kg arm.
Measure: Median (Full Range); unit: hour
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 6 | 6 | 0 | 4 | 0 | 7 | 6 | 4
hour
  Day 1 | 0.75 [0.50 to 23.92] | 0.75 [0.50 to 23.92] |  | 3.49 [0.50 to 12.00] |  | 1.00 [1.00 to 23.92] | 1.00 [0.98 to 23.92] | 1.49 [0.98 to 6.00]
  Day 12: number analyzed (Participants) | 6 | 6 | 0 | 4 | 0 | 6 | 6 | 4
  Day 12 | 0.75 [0.50 to 1.00] | 1.00 [0.50 to 4.00] |  | 1.50 [0.50 to 1.98] |  | 1.00 [1.00 to 1.50] | 1.00 [0.50 to 6.00] | 0.98 [0.50 to 2.98]

14. Secondary Outcome: Apparent Terminal Half-life
Description: Apparent Terminal Half-life (t1/2) is the time required for a given MK-5160 concentration in the plasma to decrease by 50%.
Time Frame: as for outcome 5
Population: All participants that received MK-5160, had no major protocol violations, and had t1/2 values available on Day 1 and Day 12. t1/2 was not calculated for the Glargine 0.4 U/kg and 0.6 U/kg arms. No participants were randomized to the T1DM MK-5160 64 nmol/kg or T2DM MK-5160 16 nmol/kg arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 6 | 6 | 0
hour | 20.01 (59.84) | 21.69 (27.70) |  |  |  | 13.10 (36.05) | 14.47 (16.78) |

ADVERSE EVENTS:
Time Frame: Up to 33 days
Description: All participants who received at least one dose of study drug. No participants were randomized to the T1DM MK-5160 64 nmol/kg arm or the T2DM MK-5160 16 nmol/kg arm.
Arm/Group | T1DM MK-5160 16 Nmol/kg | T1DM MK-5160 32 Nmol/kg | T1DM MK-5160 64 Nmol/kg | T1DM Glargine 0.4 U/kg | T2DM MK-5160 16 Nmol/kg | T2DM MK-5160 32 Nmol/kg | T2DM MK-5160 64 Nmol/kg | T2DM Glargine 0.6 U/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/0 | 0/4 | 0/0 | 0/7 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/0 | 0/4 | 0/0 | 0/7 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 0/0 | 4/4 | 0/0 | 7/7 | 6/6 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T1DM MK-5160 16 Nmol/kg (N=6) | T1DM MK-5160 32 Nmol/kg (N=6) | T1DM MK-5160 64 Nmol/kg (N=0) | T1DM Glargine 0.4 U/kg (N=4) | T2DM MK-5160 16 Nmol/kg (N=0) | T2DM MK-5160 32 Nmol/kg (N=7) | T2DM MK-5160 64 Nmol/kg (N=6) | T2DM Glargine 0.6 U/kg (N=4)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (7) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 3 (4) | 2 (2)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (8) | 0 (0) | 1 (2) | 1 (1) | 3 (6)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (68) | 5 (54) | 0 (0) | 4 (38) | 0 (0) | 1 (1) | 3 (7) | 2 (2)
Pseuodohypoglycaemia (Metabolism and nutrition disorders) | 2 (6) | 5 (13) | 0 (0) | 3 (6) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT03095651/Prot_SAP_000.pdf